CLINICAL TRIAL: NCT02803632
Title: Clinical and Actigraphic Profile of Young Patients Admitted for Attempted Suicide: Investigation of Disruptive Mood Dysregulation Disorder
Brief Title: Clinical and Actigraphic Profile of Young Patients Admitted for Attempted Suicide
Acronym: ACTIHUMEUR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment problem
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AOL11-DR -GUILE
Record Dates: First submitted 2016-06-09; First posted 2016-06-17 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Suicide, Attempted
Keywords: young; disruptive mood dysregulation disorder; actigraphic profile
MeSH Terms: conditions — Suicide, Attempted | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- suicide attempt (Experimental): questionnaires actigraphic recording
  Interventions: Behavioral: questionnaires; Device: actigraphic recording

INTERVENTIONS:
Behavioral: questionnaires
Device: actigraphic recording

SUMMARY:
An excess suicide-related morbidity is observed among young people in the Picardie region, as reflected by the > 100% occupation rate of the Amiens University Hospital Adolescent Medicine Unit

DETAILED DESCRIPTION:
An excess suicide-related morbidity is observed among young people in the Picardie region, as reflected by the > 100% occupation rate of the Amiens University Hospital Adolescent Medicine Unit. New approaches have been proposed to these problems that have led us to reorganize our diagnostic practices: 1) more precise characterization of suicidal behaviour by using standardized instruments such as the French version of the Columbia-Suicide Severity Rating Scale developed by Posner (C-SSRS); 2) new clinical entities, such as disruptive mood dysregulation disorder, are now proposed in international classifications (DSM 5 field trial); 3) investigations such as recording of the circadian rhythm of motor activity by actigraphy are being studied as a laboratory complement to psychiatric diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* children/adolescents admitted after a suicide attempt

Exclusion Criteria:

* severe depression
* mental retardation
* pervasive developmental disorder
* active psychotic episode,
* drug and alcohol abuse at the time of admission
* organic sleep-wake disorders (sleep-related respiratory and motor disorders, narcolepsy)
* any contraindication formulated by the clinical team
* patients not covered by French national health insurance, patients deprived of their freedom as stipulated in Article L.1121-6 of the French Public Health Code

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2013-02-06 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
The variable absence / presence of the disruptive mood dysregulation disorder (DMDD) | Day 0
  The variable absence / presence of the disruptive mood dysregulation disorder (DMDD)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc GUILE, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens
  - AP HP, Paris